CLINICAL TRIAL: NCT03313609
Title: Investigating Burnout in Intensive Care in Middle Incoming Turkey
Acronym: burnout
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Ersin Arslan Education and Training Hospital (Other Government)
Responsible Party: Principal Investigator, gulserenelay, Dr. Ersin Arslan Education and Training Hospital, Dr. Ersin Arslan Education and Training Hospital
Other Study IDs: No sponsor
Record Dates: First submitted 2017-10-14; First posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Burnout Syndrome
MeSH Terms: conditions — Burnout, Psychological | interventions — Critical Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Investigating Burnout in Intensive Care in Middle Incoming Turkey — single-group studies
  Other Names: ilhan bahar

SUMMARY:
Turkey is a developing country and its intensive care infrastructure is worse than developed countries. The staff is very busy at work. Intensive care has become a new science. We wanted to investigate burnout syndrome among physicians and other health care workers who are starting to work at a new intensive care medicine. Intensive care specialists in Turkey do not work in intensive care centers where they want. This may have a negative effect on physicians.

DETAILED DESCRIPTION:
Burnuot health practices are more common than the normal group. The data about Turkey are limited. In developing societies, there are often no protocols in intensive care. There are no teams again during intensive care. All work is done by physicians and other health workers. This may adversely affect health care workers. Intensive care science is new. The training first started in 2013. The newly graduated heavy-duty specialists can work where they do not want. The workload of the health workers working in the intensive care unit is high. We wanted to investigate burnout on healthcare workers in Turkey.

ELIGIBILITY:
Inclusion Criteria:

fellow, nursing, specialist and academics working intensive care medicine

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: working intensive care medicine
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2017-10-25 (Estimated); Study Completion 2017-11-05 (Estimated)

PRIMARY OUTCOMES:
maslach burnout inventory measure | 20 day

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Ersin Arslan Education and Training Hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No